CLINICAL TRIAL: NCT03845751
Title: EvaluatioN of High-intensity Focused Ultrasound (HIFU) Hemiablation and Short Term AndrogeN Deprivation Therapy Combination to Enhance Prostate Cancer Control for Intermediate Risk Localized Prostate Cancer: the ENHANCE Prospective Feasibility Trial.
Brief Title: EvaluatioN of HIFU Hemiablation and Short Term AndrogeN Deprivation Therapy Combination to Enhance Prostate Cancer Control.
Acronym: ENHANCE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Mutualiste Montsouris (Other)
Collaborators: University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: URO-01-2019
Record Dates: First submitted 2019-01-24; First posted 2019-02-19 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer; Androgen Deprivation Therapy
Keywords: HIFU; hemi ablation; focal therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADT protocol (Experimental): ADT protocol is administered as a single subcutaneous injection of 3-month depot of 22.5 mg of leuprolide acetate (luteinizing hormone-releasing hormone [LHRH] agonist). ADT protocol starts one month prior to the scheduled HIFU session. The intervention of the study is HIFU hemi-ablation combined with ADT.
  Interventions: Drug: HIFU hemi-ablation combined with ADT.

INTERVENTIONS:
Drug: HIFU hemi-ablation combined with ADT. — Hemi-ablation of the cancer-harbouring prostatic lobe will be carried out using HIFU energy. Short-term 3-month ADT will be administered concomitantly. Short-term ADT is administered as a single subcutaneous injection of 3-month depot of 22.5 mg of leuprolide acetate (luteinizing hormone-releasing hormone [LHRH] agonist). The ADT protocol starts within 1 month prior to the scheduled HIFU session

SUMMARY:
The current study aims to examine the hypothesis that combining the focal effects of HIFU with the systemic effects of androgen deprivation therapy might eradicate the prostatic cancer cells by targeting the 'visible' index focus (by HIFU) and the tumour surrounding microenvironment which may contain 'invisible' foci and aberrant PCa related signalling (by androgen deprivation therapy) to enhance oncological outcomes of HIFU hemi-ablation in men with localized PCa, and consequently reducing treatment failures.

DETAILED DESCRIPTION:
Prostate Cancer (PCa) is a multifocal disease in up to 90% of men with heterogeneity among different cancer foci in the same prostate gland. An index/dominant lesion has been proposed, namely the largest tumor nodule that often correlates with the highest Gleason score (GS) and, consequently, with the clinical behavior of the tumor. However, this concept is not always applicable as highest GS, largest tumor volume and extraprostatic extension may be present in different PCa foci in up to 10% of the cases.

Focal therapies (FT) for localized PCa emerged to reduce the adverse effects of radical treatments,including a30-90% for erectile dysfunction and 5-20% for incontinence and rectal toxicity, while maintaining comparable oncological efficacy. Amongst organ-sparing strategies, high-intensity focused ultrasound (HIFU) is widely used and yields promising cancer control rates and relatively low morbidity.

In our recently published prospective study of HIFU hemiablation for localized PCa with one year follow up, 25.4% of patients demonstrated PCa cores at 12 months post-treatment biopsy (Feijo et al, Eur Urol, 2016). Among them 11.5% of patients showed cancer in the contralateral untreated lobe. At 3 months, all patients were continent and 11 out of 21 preoperatively potent patients maintained adequate sexual functions. Minor adverse effects were reported in 8%, while 2.8% of patients experienced Clavien-Dindo grade-3 events.

Although FT has proven to be effective and less morbid treatment for localized PCa, an area for improvement still exists and a gap in cancer control needs to be filled by adding additional form of treatment so as to improve oncological outcomes and minimize treatment failures.

Research Rationale Previous studies have shown approximately 20% of men continue to harbour cancer at 12 months after HIFU FT for localized PCa. This finding could be in part attributed to undetectable (invisible) remote cancer foci owing to limitations of the currently available imaging and biopsy techniques and representing an appealing argument against FT.

Another point is tumor microenvironment, defined as the myriad of multiple interactions amongst tumour and surrounding cells including immune cells, stromal fibroblasts, mesenchymal stem cells and blood vessels.

It is not completely clear whether at least part of FT recurrences may be related to non-aggressive lesions taking the position of an index PCa focus and/or PCa index lesion signalling altering benign tissues behaviour.

Androgen deprivation therapy (ADT) modifies tumour microenvironment and suppresses PCa growth and progression.

Short-term ADT has been reported to increase the overall survival in men with localized intermediate- to high-risk PCa when combined with external beam radiation therapy (EBRT) or RP.

Short term ADT has been also investigated in the context of active surveillance; other trials are under way.

However, to date, there is no prospective data assessing the role of HIFU/ADT combination therapy for the treatment of localized PCa in terms of cancer control.

The current study aims to examine the hypothesis that combining the focal effects of HIFU with the systemic effects of androgen deprivation therapy might eradicate the prostatic cancer cells by targeting the 'visible' index focus (by HIFU) and the tumour surrounding microenvironment which may contain 'invisible' foci and aberrant PCa related signalling (by androgen deprivation therapy) to enhance oncological outcomes of HIFU hemi-ablation in men with localized PCa, and consequently reducing treatment failures, without significantly increasing toxicity and/or complications.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 40 and over.
* Life expectancy ≥ 10 years.
* Localized, intermediate-risk PCa (according to the most recent version of the European Association of Urology Prostate Cancer Guidelines).
* PI-RADS ≥ 3 lesions in MRI (PI-RADS v2.1).
* Unilateral (unifocal or multifocal) PCa or bilateral disease allowing unilateral GS 3+3 up to 1mm in the non-treated side.
* Histopathologically verified PCa by any mpMRI-targeted prostate biopsy (3 cores per each target lesion + 12 random cores performed).
* Any Gleason score 7 (3 + 4) (ISUP2).
* Prostate specific antigen (PSA) ≤15 ng/ml.
* Clinical stage T1c-T2b (based on MRI and/or rectal examination).
* Absence of lymph node and distant metastases.
* Prostate volume ≤ 60 ml. Patient with prostate volume between 40 ml and 60 ml could be included only if lesion is located in posterior zone of the prostate.
* Treatment-naive patients (received no previous treatments for PCa, apart from active surveillance).
* World Health Organization (WHO) performance status of grade 0-2.
* Men who are sexually active with women of chidbearing potential must use a highly effective method of contraception prior the first administration of hormonal therapy and must agree to continue using such precautions for 130 days after the final administration of the treatment.
* Having signed a written informed consent form.

Exclusion Criteria:

* Men under the age of 40.
* Life expectancy less than 10 years.
* Any Gleason score ≤6 (3 + 3) (ISUP1).
* Any Gleason score≥ 7 (4+3) (ISUP3).
* PI-RADS < 3 lesions in MRI (PI-RADS v2.1).
* Apex lesions may ≥ 10 mm away from the urethral sphincter.
* PSA >15 ng/ml.
* Clinical stage > cT2b (based on MRI and rectal examination).
* Evidence of extra-prostatic extension or seminal vesicle invasion.
* Evidence of lymph node or distant metastases.
* Prostate volume > 40 ml when lesion is located in the anterior zone of the prostate.
* Prostatic calcifications or cysts whose location may interfere with effective delivery of HIFU energy.
* Metal implants/stents in the urethra.
* Active urinary tract infection.
* Men who have previously received any form of PCa treatment (e.g. external beam radiation therapy (EBRT), brachytherapy, HIFU, cryosurgery, thermal or microwave therapy and/or hormonal therapy).
* Patient treated with 5 α-reductase inhibitors in the previous 3 months and during the study.
* Men who have undergone surgery for benign prostatic hyperplasia in the previous 6 months; i.e. a transurethral resection of the prostate (TURP), holmium laser enucleation (HOLEP), greenlight laser vaporization, others.
* Men with an inability to tolerate a transrectal ultrasound probe or have undergone prior significant rectal surgery preventing insertion of transrectal HIFU probe.
* Men unable to have MRI scanning (e.g. men with severe claustrophobia, permanent cardiac pacemaker or metallic implant which may likely contribute to significant image artefacts).
* Men with renal impairment and a glomerular filtration rate (GFR) of <35 ml/min (unable to tolerate Gadolinium dynamic contrast enhanced MRI).
* WHO performance status of grade 3-4 / men unfit for surgery.
* Hypersensitivity to leuprorelin acetate, to other GnRH agonists or to any of the excipients.
* Men with congenital long QT syndrome, congestive heart failure, frequent electrolyte abnormalities, or taking drugs known to prolong the QT interval.
* Patients who previously underwent orchidectomy.
* Language barriers that might hinder the communications, understanding of written and verbal information about the trial, consenting process, or completing the questionnaires.
* Men refusing to sign an informed consent to participate in the trial.
* Men with relative and/or absolute contraindications to androgen deprivation therapy.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Oncological outcome | 12 months after the HIFU session
  Number of treatment failures determined after prostatic biopsy and defined as:
  * Any Gleason pattern ≥4.
  * Any Gleason score ≥7.

SECONDARY OUTCOMES:
Urinary continence | 1, 3, 6 and 12 months post-treatment
  Rate of men maintaining continence and becoming incontinent after treatment. Continence is defined as >0pad/day being used. Incontinence is defined conversely.
Urinary continence variation | at 1, 3, 6 and 12 months post-treatment
  Variation of ICSmale SF score in incontinence domains (international continence society male short form questionnaire - incontinence domain is composed by six questions going from 0 (total continence) to 24 (severe incontinence).
Urinary continence proportion | 1,3, 6, and 12 months post-treatment
  Variation in continence category according to the number of pads used/day due to continence problems compared to baseline. Categories will be (full continence= 0 pads/day or security pad, mild incontinence =1pad/day, moderate incontinence= 2pads/day, severe incontinence >2pads/day).
Urinary voiding function variation | 1,3, 6, and 12 months post-treatment
  Urinary voiding function variation (compared to baseline) assessing changes of the IPSS (International Prostatic Symptoms Score).
  The IPSS score measures if the subject has significant problems/symptoms in passing the urine/voiding the bladder. The scale goes from 0 (no symptoms or bother) to 35 (extremely severe symptoms).
Erectile function | 1, 3, 6 and 12 months post-treatment
  Rate of men maintaining potency after treatment. Erectile function changes will be assessed using the IIEF-5 and considering potency as IIEF-5 ≥22 without need of any medication (PDE-5 inhibitors and/or others).
Erectile function variation | at 1, 3, 6 and 12 months post-treatment
  Erectile function as compared to baseline using:
  * IIEF-5 score changes at different time points post-treatment, as compared to baseline.
  * Proportion of men who are potent at baseline and then sustain erectile dysfunction, at 12 months. Potency is defined as an IIEF score ≥22 without requiring any medication.
Ejaculatory function | 1, 3, 6 and 12 months post-treatment as compared to baseline.
  Ejaculatory function compared to baseline using MSHQ-EjD questionary at time points post-treatment.
Treatment toxicity and complications | 12 months
  Rate of men experiencing treatment related complications and toxicity. Surgical complications will be graded using the Clavien-Dindo classification. Treatment related toxicity and adverse events will be graded using the Common Terminology Criteria for reporting Adverse Events (CTCAE v5).
Additional treatment due to recurrent or persistent prostate cancer | 12 months
  Rate (%) of men needing to undergo further prostate cancer active treatment due to treatment failure due to biochemical recurrence according to the Phoenix criteria and biopsy proving persistence/recurrence of clinically significant PCa (defined as previously described - see Oncological outcome).
Quality of life variation | 1, 3, 6 and 12 months post-treatment.
  Evolution of quality of life compared to baseline at timepoints post-treatment using EQ-5D-5L questionary.
PSA variation | at 1, 3, 6, and 12 months post-treatment, as compared to baseline.
  Serum free and total PSA levels changes
Testosterone variation | at 1, 3, 6, and 12 months post-treatment, as compared to baseline
  Serum Testosterone levels changes .

CONTACTS AND LOCATIONS:
Overall Officials: Lara RODRIGUEZ-SANCHEZ, Doctor, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Institut Mutualiste Montsouris, Paris, France

IPD SHARING:
Plan to Share IPD: No